CLINICAL TRIAL: NCT05476484
Title: Comparative Real World Effectiveness of SQ Sublingual Immunotherapy (SLIT)-Tablets vs. Controls in Allergic Rhinitis and Asthma - Outcomes From a Multinational Register Study
Brief Title: Comparative Real World Effectiveness of SQ Sublingual Immunotherapy (SLIT)-Tablets vs. Controls in Allergic Rhinitis and Asthma
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: ALK-Abelló A/S (Industry)
Collaborators: Quantify Research (Unknown)
Responsible Party: Sponsor
Other Study IDs: NI-X-05
Record Dates: First submitted 2022-06-29; First posted 2022-07-27 (Actual); Last update posted 2023-08-02 (Actual); Status verified 2023-07

CONDITIONS: Allergy; Allergic Rhinitis; Asthma
Keywords: Allergy immunotherapy; Sublingual immunotherapy (SLIT)-tablets; Grass; House dust mite; Retrospective cohort study
MeSH Terms: conditions — Hypersensitivity; Rhinitis, Allergic; Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Allergic rhinitis patients with and without asthma treated with SQ SLIT-tablet
  Interventions: Drug: SQ SLIT-tablet
- Allergic rhinitis patients with and without asthma not treated with SQ SLIT-tablet

INTERVENTIONS:
Drug: SQ SLIT-tablet — SQ grass SLIT-tablet and/or SQ house dust mite SLIT-tablet
  Groups: Allergic rhinitis patients with and without asthma treated with SQ SLIT-tablet

SUMMARY:
To assess the impact of SQ SLIT-tablets (SQ Grass SLIT-tablet and SQ HDM SLIT-tablet) in Danish and Swedish allergic rhinitis (AR) patients, with or without asthma, between 2007-2020.

DETAILED DESCRIPTION:
Allergic rhinitis (AR) is an inflammatory disorder, characterised by pruritus, sneezing, rhinorrhoea, and nasal congestion. It is one of the most common disorders worldwide, with an estimated global prevalence of 10-30%. AR is a chronic and progressive disease, as the underlying respiratory allergy can progress into allergic asthma. The prevalence of asthma in patients with AR is high and estimated between 10-40%. The presence of AR commonly exacerbates asthma, increasing the risk of asthma exacerbations, emergency visits and hospitalisations for asthma.

Recently, the high-quality retrospective cohort REACT study (ClinicalTrial.gov: NCT04125888) found that allergy immunotherapy (AIT) was associated with long-term reduction in AR medication use as well as significant reductions in both controller and reliever asthma medication and concurrent lower risk of asthma exacerbation and pneumonia in subjects with pre-existing asthma. The SQ sublingual immunotherapy (SLIT)-tablets have robust evidence from randomised controlled trials (RCTs), but real-world evidence (RWE) is needed to complement the findings from RCTs by looking at e.g. longer time horizons and broader patient populations. As the REACT study was not designed to specifically look at evidence-based AIT treatments like the SQ SLIT-tablets, the real-world effectiveness of SQ SLIT tablets remain to be further elucidated.

ELIGIBILITY:
Inclusion Criteria:

AR-patients identified by dispensations of prescribed AR medications and/or ICD10-codes of AR in specialty care

For the SQ SLIT-tablet cohort:

- at least 2 dispensings within 365 days of SQ SLIT-tablets (ATC: V01AA02 and V01AA03)

For the control cohort:

- unexposed subjects will be identified from the study population of AR-patients that may be eligible to receive SQ SLIT-tablets, but have not dispensed a prescription of SQ SLIT-tablets during the index year of the case or prior to that year

Exclusion Criteria:

- allergy immunotherapy treatment with grass or HDM allergens prior to the index event

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: AR-patients identified by dispensations of prescribed AR medications and/or ICD10-codes of AR in specialty care
Sampling Method: Probability Sample
Enrollment: 49844 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Symptom-relieving medication use for allergic rhinitis | From pre-index to follow-up year(s), assessed from 2005 and up to 2021
  Overall number of prescriptions and by individual drug classes

SECONDARY OUTCOMES:
Medication use for asthma | From pre-index to follow-up year(s), assessed from 2005 and up to 2021
  Overall number of prescriptions and by individual drug classes
Asthma disease severity assessed by reliever and controller medication prescriptions and hospitalisations due to asthma | From pre-index to follow-up year(s), assessed from 2005 and up to 2021
Lower airway infections assessed by prescriptions of antibiotics and diagnosis codes for pneumonia | From pre-index to follow-up year(s), assessed from 2005 and up to 2021

OTHER OUTCOMES:
Health care resource utilisation assessed by ambulatory care visits | From pre-index to follow-up year(s), assessed from 2005 and up to 2021
Health care resource utilisation assessed by hospitalisations | From pre-index to follow-up year(s), assessed from 2005 and up to 2021
Health care resource utilisation assessed by cost | From pre-index to follow-up year(s), assessed from 2005 and up to 2021

CONTACTS AND LOCATIONS:
Overall Officials: Julie F Rask Larsen, MD PhD, Study Director — ALK
Locations (1):
- ALK, Hørsholm, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No